CLINICAL TRIAL: NCT03803436
Title: Improving Outcome of Selected Patients With Non-resectable Hepatic Metastases From Colo-rectal Cancer With Liver Transplantation: a Prospective Parallel Trial
Brief Title: Improving Outcome of Selected Patients With Non-resectable Hepatic Metastases From Colo-rectal Cancer With Liver Transplantation
Acronym: COLT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other); Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 108/18
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Liver Metastases; Colorectal Cancer Metastatic; Liver Neoplasm; Neoplasms
Keywords: Liver Transplant; Colorectal Cancer; Chemotherapy; Metastasis
MeSH Terms: conditions — Liver Neoplasms; Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis | interventions — Liver Transplantation; Drug Therapy

STUDY DESIGN:
Intervention Model Description: The study will compare survival in the population of patients enrolled in the COLT trial with the OS in the COLT-eligible population enrolled in the parallel TRIPLETE trial conducted by the GONO Group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): Liver transplant
  Interventions: Procedure: Liver transplant
- Parallel arm (Active Comparator): Chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Liver transplant — Liver transplant from cadaveric donors
  Arms: Study arm
Drug: Chemotherapy — mFOLFOX
  Arms: Parallel arm
Drug: Chemotherapy — Panitumumab
  Arms: Parallel arm

SUMMARY:
The COLT trial is an investigator-driven, multicenter, non-randomized, open-label, controlled, prospective, parallel trial, aimed at assessing the efficacy (in terms of overall survival: OS) of liver transplantation (LT) in liver-only CRC metastases, compared with a matched cohort of patients bearing the same tumor characteristics, collected during the same time period and included in a phase III Italian RCT on triplet chemotherapy+antiEGFR

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-mucinous colon adenocarcinoma.
* Primary tumor as pT1-3, pN0 or pN1 (metastases in < 4 regional lymph nodes), confirmed R0 resection.
* RAS and BRAF wild-type & MSS molecular status as per local testing.
* Liver metastases not eligible for curative liver resection
* Objective response according to RECIST 1.1 to first-line treatment, with sustained response for at least 4 months, OR disease control (CR+PR+SD) during second-line treatment for at least 4 months.
* A maximum of two prior chemotherapy treatment lines.
* Performance status, ECOG 0.
* Satisfactory blood tests Hb >10g/dl, neutrophils >1.0 (after any G-CSF), TRC >75, Bilirubin<2 x upper normal level, AST, ALT<5 x upper normal level, creatinine <1.25 x upper normal level.
* CEA<50 ng/ml

Exclusion Criteria:

* Hereditary CRC syndromes including FAP and Lynch syndrome.
* Prior extra hepatic metastatic disease or primary tumor local relapse.
* Extra-peritoneal cancers (rectum).
* Other malignancies in the previous 5 years
* Active intra-venous or alcohol abusers
* HIV infection

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  Time from enrolement to either death or censoring

SECONDARY OUTCOMES:
Progression Free Survival | 5 years
  Time from enrolement to either progression or censoring
Complications rate | 90 days after liver transplant
  Complications according to Dindo Clavien Classification

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Mazzaferro, MD, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori di Milano
Locations (12):
- Italy (12):
  - SOD Clinica di Chirurgia Epatobiliare, Pancreatica e dei Trapianti e SC di Oncologia Medica, Ospedali Riuniti di Ancona, Ancona
  - ASST Papa Giovanni XXIII, Bergamo
  - Chirurgia EBP e dei Trapianti di Fegato e SC di Oncologia Medica, Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Istituto NAzionale Tumori di Milano, Milan
  - Ospedale Maggiore di Milano Policlinico, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione (ISMETT), Palermo
  - GONO Group (Gruppo Oncologico Nord Ovest) TRIPLETE Trial Coordination, Pisa
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma
  - Ospedale Universitario Molinette S. Giovanni Battista di Torino, Torino
  - Centro Trapianti di Fegato e SC di Oncologia Medica, A.S.U. Integrata di Udine, Udine
  - Centro Trapianti di Fegato e SC di Oncologia Medica, A.O.U. Integrata di Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sposito C, Pietrantonio F, Maspero M, Di Benedetto F, Vivarelli M, Tisone G, De Carlis L, Romagnoli R, Gruttadauria S, Colledan M, Agnes S, Ettorre G, Baccarani U, Torzilli G, Di Sandro S, Pinelli D, Caccamo L, Sartore Bianchi A, Spreafico C, Torri V, Mazzaferro V. Improving Outcome of Selected Patients With Non-Resectable Hepatic Metastases From Colorectal Cancer With Liver Transplantation: A Prospective Parallel Trial (COLT trial). Clin Colorectal Cancer. 2023 Jun;22(2):250-255. doi: 10.1016/j.clcc.2023.01.003. Epub 2023 Feb 3. PMID 36822922